CLINICAL TRIAL: NCT03435393
Title: Ripple-Mapping for the Detection of Long Duration Action Potential Areas in Patients With Brugada Syndrome
Brief Title: Ripple Mapping for Epicardial Mapping of Brugada Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College London Hospitals (Other)
Responsible Party: Principal Investigator, Rui Providência, Honorary Consultant, MD PhD, University College London Hospitals
Other Study IDs: Barts_Brugada
Record Dates: First submitted 2018-02-09; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Brugada Syndrome
MeSH Terms: conditions — Brugada Syndrome | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Catheter ablation — Mapping of the epicardium and ablating areas of long fractionated potentials

SUMMARY:
Whether a mapping algorithm "Ripple-mapping" is able to rapidly identify the areas of long-duration multicomponent electrograms which constitute the targets for ablation for an automated strategy remains to be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Brugada syndrome patients requiring ablation

Exclusion Criteria:

* Patients not able to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Brugada syndrome and an episode of ventricular tachycardia
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Eradication of Brugada syndrome pattern | 24h post procedure
  Disappearance of type 1 Brugada pattern on post-procedure ECG

SECONDARY OUTCOMES:
Freedom from ventricular arrhythmias | 12 months post-procedure
  No documentation of sustained ventricular tachycardia or ventricular fibrillation

CONTACTS AND LOCATIONS:
Locations (3):
- Instituto do Coracao, São Paulo, Brazil
- Hospital de Santa Cruz, Lisbon, Portugal
- St Bartholomew's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Patient data will be anonymised